CLINICAL TRIAL: NCT01805219
Title: Assessment of Human Locomotion and Energy Expenditure Using Global Positioning Satellite and Accelerometry
Brief Title: Global Positioning Satellite and Accelerometry to Assess Human Locomotion (ACTI GPS)
Acronym: ActiGPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Collaborators: École Normale Supérieure de Cachan (Other); Institut de Formation en Education Physique et en Sport d'Angers/Les Ponts de Cé (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2012-A01411-42
Record Dates: First submitted 2013-02-18; First posted 2013-03-06 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- healthy subjects
  Interventions: Other: GPS and accelerometer recording (s) during exercises

INTERVENTIONS:
Other: GPS and accelerometer recording (s) during exercises

SUMMARY:
The aim of the study is to validate the association of the GPS and accelerometer tools in order to assess the humain locomotion during exercises.

The hypotheses are:

1. GPS and accelerometer together can assess the human locomotion
2. GPS and accelerometer together can assess the energy expenditure during exercises

DETAILED DESCRIPTION:
The assessment of the physical activity (PA) and the energy expenditure (EE) is very important to estimate the morbi-mortality. However, each of these tools has its advantages and disadvantages but none of them provides a measure of all components dimensions that characterize the associated PA and EE. The current scientific prospects for measurement of PA tend to associate several measuring devices. To date, these perspectives are facilitated by technological developments and miniaturization of various devices. Thus, the purpose of the study is to evaluate wether GPS associated with accelerometer are able to assess the humain locomotion and energy expenditure during exercises.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18
* Informed consent of the participant
* Able to understand the protocol of the study
* Register to the social health insurance
* No exercise limitation

Exclusion Criteria:

* No informed consent of the participant
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2016-06-08 (Actual)

PRIMARY OUTCOMES:
Defining optimal analysis parameter to accurately detect walking from stopping periods | up to 1 week
  Predefined walking protocols will be recorded and the subjects asked to follow recorded procedures.
  Detection performance of walking and resting bouts (expressed by the percentage accuracy in the detection of walking and resting bouts actually performed) for: i) GPS alone; ii) Accelerometer alone; iii) both GPS and accelerometer

SECONDARY OUTCOMES:
Defining optimal analysis parameter to accurately detect speed and distance of periods of walking | up to 1 week
  Predefined walking protocols will be recorded and the subjects asked to follow recorded procedures at a defined walking pace.
  Accuracy of speed and distance estimations (expressed by the typical error of estimate and the coefficient of variation) from: i) GPS alone; ii) Accelerometer alone; iii) both GPS and accelerometer.

OTHER OUTCOMES:
Determine the accuraccy of GPS and acceleropmetry to estimate energy expediture in healthy volunteers | up to 1 week
  Recording of VO2 real time with a portable analyser in parallel to GPS and accelerometry.
  Prediction (determined by the coefficient of determination from linear regression) of energy expenditure during level and grade outdoor walking and running from: i) GPS alone; ii) Accelerometer alone; iii) both GPS and accelerometer.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Angers, France

REFERENCES:
- [Derived] de Mullenheim PY, Dumond R, Gernigon M, Mahe G, Lavenu A, Bickert S, Prioux J, Noury-Desvaux B, Le Faucheur A. Predicting metabolic rate during level and uphill outdoor walking using a low-cost GPS receiver. J Appl Physiol (1985). 2016 Aug 1;121(2):577-88. doi: 10.1152/japplphysiol.00224.2016. Epub 2016 Jul 8. PMID 27402559